CLINICAL TRIAL: NCT07105046
Title: Facilitators and Barriers to Cancer Treatment Among Texas Residents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-0697; NCI-2025-05584 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic; Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-structured Interview (Experimental): Participants will be recruited through the Texas Cancer Registry (TCR).
  Interventions: Other: Focus Groups
- Online Focus Group (Experimental): Participants will be recruited through the Texas Cancer Registry (TCR).
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — A 30 to 45-minute in-depth semi-structured interview by phone will be administer, following a semi-structured interview guide.
  Arms: Online Focus Group
Other: Focus Groups — 45 to 60 minutes video conference
  Arms: Semi-structured Interview

SUMMARY:
This trial uses semi-structured interviews and focus groups to determine facilitators and barriers of receiving timely cancer treatment among multiple cancers, across multiple insurance types, throughout Texas

DETAILED DESCRIPTION:
Primary Objectives:

Aim 1: To comprehensively assess barriers to and facilitators of receiving timely cancer treatment, via in-depth telephone interviews among a purposive sample of Texas patients with Stage I-IV breast, colorectal, lung, and prostate cancer and diverse backgrounds.

Aim 2: To generate consensus on barriers and facilitators, as well as their relative importance, via focus groups, among carefully selected Texas patients with Stage I-IV breast, colorectal, lung and prostate cancer and diverse backgrounds,

ELIGIBILITY:
Inclusion Criteria:

Aims 1 and 2

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Verbal consent will be obtained
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Males and females; Age ≥ 18 years old
* Documented diagnosis of breast, colorectal, lung, and prostate cancer patients, stage I-IV
* Either English or Spanish-speaking

Exclusion Criteria:

Aims 1 and 2

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patients who are cognitively impaired
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: John Lin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org